CLINICAL TRIAL: NCT03363867
Title: BEACON - A Phase II Study of Bevacizumab, Atezolizumab and Cobimetinib in Patients With Recurrent Platinum Resistant High Grade Serous Ovarian Cancer
Brief Title: BEACON - ABC in Recurrent Platinum Resistant HGSOC
Acronym: BEACON
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Peter MacCallum Cancer Centre, Australia (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BEACON
Record Dates: First submitted 2017-11-28; First posted 2017-12-06 (Actual); Last update posted 2023-08-07 (Actual); Status verified 2023-08

CONDITIONS: Ovarian Cancer; Fallopian Tube Cancer; Primary Peritoneal Carcinoma
Keywords: High grade serous; Platinum resistant; Recurrent ovarian cancer
MeSH Terms: conditions — Ovarian Neoplasms; Fallopian Tube Neoplasms | interventions — atezolizumab; Bevacizumab; cobimetinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Atezolizumab, Bevacizumab and Cobimetinib (ABC) (Experimental)
  Interventions: Drug: Atezolizumab; Drug: Bevacizumab; Drug: Cobimetinib

INTERVENTIONS:
Drug: Atezolizumab — 840mg every 2 weeks (i.e. Day 1 and Day 15 of each 28 day cycle) via intravenous infusion from Cycle 2 onwards.
  Other Names: Tecentriq
Drug: Bevacizumab — 5mg/kg every 2 weeks (i.e. Day 1 and Day 15 of each 28 day cycle) via intravenous infusion.
  Other Names: Avastin
Drug: Cobimetinib — 60mg per day, every day for 21 days (i.e. Day 1 to Day 21 of each 28 day cycle)
  Other Names: Cotellic

SUMMARY:
Epithelial ovarian cancer (EOC) is the ninth most common cause of cancer in Australian women, with an estimated 1500 new diagnoses in Australia in 2015, and remains the seventh most common cause of cancer death in Australian women. High grade serous ovarian cancer (HGSC) is the most common form of Epithelial Ovarian Cancer, and accounts for the most deaths due to a gynaecological cancer.

The majority of women diagnosed with High Grade Serous Ovarian Cancer present with advanced disease, and are typically managed with a combination of cytoreductive surgery and platinum-based chemotherapy. Despite initial good response rates to chemotherapy, High Grade Serous Ovarian Cancer recurs in up to 70% of patients who present with Stage III/IV disease.

The purpose of this research project is to test how safe and effective the combination treatment of cobimetinib, bevacizumab and atezolizumab is as a treatment for patients with platinum resistant or refractory high grade serous ovarian, fallopian tube or peritoneal cancer.

Cobimetinib is a drug that blocks a protein called Mitogen-activated protein kinase (MEK). MEK proteins are involved in the multiplication of cancer cells. By binding to the MEK protein, cobimetinib may help to stop the growth of your cancer cells.

Bevacizumab is an antibody (a type of protein produced by the immune system) that is specifically designed to block a protein called Vascular Endothelial Growth Factor (VEGF). VEGF is a protein that can increase the growth of tumour cells and binding to VEGF may help to stop the growth of tumours.

Atezolizumab is a type of drug called a Programmed Cell Death Protein 1 (PD-L1) inhibitor. PD-L1 binds to PD-1 which is a type of protein found on the surface of cells in your body's immune system, and it controls the ability of your body's natural immune response to trigger the death of tumour cells. Tumour cells can hide from the immune system by using PD-L1, which stops your immune system from triggering tumour cell death.

Atezolizumab is a drug designed to block this PD-1/PD-L1 interaction by binding to PD-L1 so that PD-1 cannot bind to it and stops it from turning off your immune cells. This helps your immune system to recognise and destroy tumour cells. In turn, this potentially can stop or reverse the growth of your cancer.

Cobimetinib, bevacizumab and atezolizumab have been used alone or in combination in the treatment of many other cancers. Each of them are individually licensed for the treatment of cancers such as advanced melanoma, non-small cell lung cancer, and bladder cancer in Australia. However, this treatment combination is experimental and is not approved to treat ovarian, fallopian tube or peritoneal cancers in any country.

ELIGIBILITY:
Inclusion Criteria:

* Patient has provided written informed consent
* Able to comply with the study protocol and follow-up procedures, in the investigator's judgement
* Female patients aged ≥ 18 years at screening
* Patients with a histological diagnosis of invasive high grade serous ovarian carcinoma (HGSC) including fallopian tube and primary peritoneal cancers, as defined by histological diagnosis and immunohistochemistry profile consistent with high grade serous cancer:

  1. Other histologies including clear cell, mucinous and carcinosarcomas are excluded.
  2. Mixed histologies are allowed provided that >80% of the primary tumour is high grade serous based on diagnostic pathology review and immunohistochemistry profile consistent with high grade serous (i.e. positive for WT1, PAX8 and P53)
* Platinum resistant or refractory recurrent disease defined by GCIG CA-125 criteria or RECIST v1.1 disease progression on or within 6 months of last platinum-based chemotherapy.
* Disease that is measurable according to RECIST 1.1 and amenable to biopsy (note that lesions intended to be biopsied should not be target lesions).
* Eastern Cooperative Oncology Group performance status of 0 or 1
* Life expectancy greater than 3 months
* Adequate hematologic and organ function, defined by the following laboratory results obtained within 7 days prior to registration

  1. WBC ≥ 2.5 x 109/L
  2. Hb ≥ 9 gm/dl
  3. ANC ≥1.5 x 109/L
  4. Platelet count ≥ 100 x 109/L
  5. Creatinine clearance ≥ 30mL/min (via Cockcroft-Gault)
  6. Albumin ≥2.5 g/dL
  7. Serum bilirubin ≤ 1.5 the upper limit of normal (ULN); patients with known Gilbert's disease may have a bilirubin ≤ 3.0 x ULN
  8. INR and PTT ≤ 1.5 x ULN; amylase and lipase ≤1.5x ULN
  9. AST, ALT, and alkaline phosphatase (ALP) ≤3 x ULN
* Absence of clinically significant proteinuria as demonstrated by urine dipstick ≤ 1+ or < 1.0g of protein in a 24-hour urine collection
* Patients with ≥2+ protein on dipstick analysis at baseline must undergo a 24-hour urine collection for protein and will remain eligible if <1.0g of protein is detected within 2 weeks of randomisation
* Negative test results for Viral Hepatitis:
* Negative hepatitis B surface antigen (HBsAg) test at screening
* Negative total hepatitis B core antibody (HBcAb) test at screening, or positive total HBcAb test followed by a negative hepatitis B virus (HBV) DNA test at screenin.The HBV DNA test will be performed only for patients who have a positive total HBcAb test.
* Negative hepatitis C virus (HCV) antibody test at screening, or positive HCV antibody test followed by a negative HCV RNA test at screening.The HCV RNA test will be performed only for patients who have a positive HCV antibody test.
* Female participants must be postmenopausal (≥ 12 months of non-therapy-induced amenorrhoea) or surgically sterile (absence of ovaries and/or uterus, or who received therapeutic radiation to the pelvis) or otherwise have a negative serum pregnancy test within 14 days of the first study treatment and agree to abstain from heterosexual intercourse or use two effective contraceptive methods that result in a failure rate of <1% per year during the whole treatment period of the study and for at least 3 months (if the last study dose contained cobimetinib), 5 months (if the last study dose contained atezolizumab) or 6 months (if the last study dose contained bevacizumab) after the last dose of study treatment. Women must refrain from donating eggs during this same period.
* Patients must have recovered to ≤ grade 1 from their treatment-related AE with the exception of alopecia.
* Has consented to the use of their collected fresh tumour biopsies, archival FFPE specimen, ascites and peripheral blood samples as detailed in the protocol for translational research, including but not limited to DNA, RNA and protein based biomarker detection.

Exclusion Criteria:

* Prior treatment with CD137 agonists or immune checkpoint blockage therapies, anti programmed death-1, anti-program death-ligand 1, MEK inhibitor. Prior treatment with bevacizumab is allowed, provided a >6 month treatment free interval from the last previous dose of bevacizumab to registration.
* Treatment with systemic immunosuppressive medications, including but not limited to corticosteroids, cyclophosphamide, azathioprine, cyclosporine, methotrexate, thalidomide and anti-tumour necrosis factor (TNF) agents within 2 weeks prior to randomization, or anticipated requirement for systemic immunosuppressive medications during the trial
* Patient has had surgical procedures or significant traumatic injury within 60 days prior to registration, or it is anticipated that they will require major surgical procedures during the course of the study.
* Patients at high risk of bowel perforation or fistula
* History of bowel obstruction, including sub- occlusive disease, related to the underlying disease and history of abdominal fistula, gastrointestinal perforation or intra-abdominal abscess.
* History of colonic anastamosis
* Clinical symptoms of recent bowel obstruction or paralytic ileus, but excluding postoperative, or evidence of recto-sigmoid involvement by pelvic examination or bowel involvement on CT scan.
* Prior treatment with Hyperthermic intraperitoneal chemotherapy (HIPEC)
* Prior whole abdominal or pelvic radiotherapy
* Untreated CNS metastases. Treatment of brain metastases, either by surgical or radiation techniques, must have been completed at least 4 weeks prior to registration. Prior to registration, there are no signs of progression or hemorrhage of treated CNS metastases, eg. by MRI Brain. No ongoing need for corticosteroid treatment (anticonvulsants are allowed)
* Treatment with any investigational agent or approved therapy within 28 days or two investigational agent half-lives (whichever is longer) prior to registration.
* Malignancies other than ovarian cancer within 5 years prior to registration (or within 3 years prior to registration, provided probability of recurrence is <10%) with the exception of adequately treated carcinoma in situ of the cervix, basal or squamous cell skin cancer, melanoma in situ, and ductal carcinoma in situ treated surgically with curative intent.
* Prior radiation therapy within 28 days prior to registration and/or persistence of radiation-related adverse effects.
* Spinal cord compression not definitively treated with surgery and/or radiation.
* Uncontrolled pleural effusion, pericardial effusion, or ascites requiring recurrent drainage procedures.
* History of autoimmune disease including but not limited to myasthenia gravis, myositis, autoimmune hepatitis, systemic lupus erythematosus, rheumatoid arthritis, inflammatory bowel disease, vascular thrombosis associated with antiphospholipid syndrome, Wegener's granulomatosis, Sjögren's syndrome, Guillain-Barre syndrome, multiple sclerosis, vasculitis, or glomerulonephritis
* Patients must not receive live, attenuated influenza vaccine (e.g., FluMist) within 4 weeks prior to registration or at any time during the study and for at least 5 months after the last dose of study drug.
* Active infection requiring IV antibiotics at screening
* Patients with known HIV infection or a history of positive tests for HIV/AIDS
* Current or recent (within 10 days of registration) use of acetylsalicylic acid (> 325 mg/day), clopidogrel (>75 mg/day) or thrombolytic agents for therapeutic purposes
* Patient has taken the following foods/supplements within 7 days prior to registration: St John's wort or hyperforin (potent CYP3A4 enzyme inducer) or Grapefruit juice (potent CYP3A4 enzyme inhibitor)
* History of severe allergic, anaphylactic, or other hypersensitivity reactions to chimeric or humanized antibodies or fusion proteins
* Known hypersensitivity or allergy to biopharmaceuticals produced in Chinese hamster ovary cells or any components of cobimetinib, atezolizumab, or bevacizumab formulations
* History of clinically significant cardiac or pulmonary dysfunction including the following; Inadequately controlled hypertension (that is defined as systolic blood pressure > 140 mmHg and/or diastolic blood pressure > 90 mmHg that is treated or untreated) or History of myocardial infarction within 6 months prior to first dose of study drug in Cycle 1
* Prior history of hypertensive crisis or hypertensive encephalopathy
* Significant vascular disease (e.g. aortic aneurysm requiring surgical repair or recent arterial thrombosis) within 6 months of registration
* History of stroke or transient ischemic attack within 6 months prior of registration
* Patient has has a serious non-healing wound, active ulcer or untreated bone fracture
* History of hemoptysis (>½ teaspoon of bright red blood per episode), or any other serious haemorrhage or at risk of bleeding (gastrointestinal history of bleeds, gastrointestinal ulcers, etc.)
* History or evidence of inherited bleeding diathesis or significant coagulopathy at risk of bleeding
* Any previous venous thromboembolism ≥ Grade 3
* Left ventricular ejection fraction below institutional lower limit of normal
* Uncontrolled serious medical or psychiatric illness
* Uncontrolled tumour pain
* History of idiopathic pulmonary fibrosis, organizing pneumonia (e.g., bronchiolitis obliterans), drug-induced pneumonitis, idiopathic pneumonitis, or evidence of active pneumonitis on screening chest CT scan
* History or evidence of retinal pathology on ophthalmologic examination that is considered a risk factor for neurosensory retinal detachment/central serous chorioretinopathy, retinal vein occlusion or neovascular macular degeneration.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Female patients with high grade serous ovarian carcinoma.
Enrollment: 30 (Actual)
Dates: Start 2018-07-10 (Actual); Primary Completion 2024-02-28 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Overall Response Rate as assessed by RECIST 1.1. | Assessed at 24 weeks after commencing treatment.

SECONDARY OUTCOMES:
The frequency and severity of adverse events with the combination treatment as assessed by CTCAE v4.03. | Through study completion, on average 12 months.
Progression free survival as assessed by RECIST 1.1. | Through study completion, on average 6 months.
Best overall response rate as assessed by RECIST 1.1. | Through study completion, on average 12 months.
Immune related tumour response rate according to iRECIST. | Through study completion, on average 6 months.
Immune related disease control rate according to iRECIST. | Assessed at 6 months after commencing treatment.
Best overall response rate as assessed by GCIG CA-125 criteria. | Through study completion, on average 12 months.

CONTACTS AND LOCATIONS:
Overall Officials: George Au-Yeung, Principal Investigator — Peter MacCallum Cancer Centre, Australia
Locations (1):
- Peter MacCallum Cancer Centre, Melbourne, Victoria, Australia